CLINICAL TRIAL: NCT06359509
Title: A Phase І Study of BCMA-targeted Chimeric Antigen Receptor T Cell (SYS6020) Injection in Relapsed or Refractory Multiple Myeloma
Brief Title: Study of SYS6020 in BCMA-positive Multiple Myeloma
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, MEI HENG, Proferssor Cheif Doctor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYS6020-001
Record Dates: First submitted 2024-03-27; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SYS6020 (Experimental): Low, medium and high doses of SYS6020 will be given.
  Interventions: Biological: BCMA Targeted CAR T-cells

INTERVENTIONS:
Biological: BCMA Targeted CAR T-cells — Each patient will receive BCMA Targeted CAR T-cells by intravenous infusion.

SUMMARY:
This is a multi-center, phase I trial that studies the efficacy and recommended dose of BCMA CART cells in treating patients with BCMA-positive multiple myeloma (MM) that have not respond or relapsed after chemotherapy. B-cell maturation antigen (BCMA), a cell surface protein expressed on malignant plasma cell, has emerged as a very selective antigen to be targeted in novel immunotherapy for MM.

ELIGIBILITY:
Inclusion Criteria:

* 1. ≥ 18 years of age at the time of signing informed consent;
* 2. Cytology or tissue biopsy meets diagnostic criteria for multiple myeloma (according to IMWG criteria);
* 3. Bone marrow specimens confirmed positive BCMA expression in plasma cells and myeloma cells by immunohistochemistry or flow cytometry (>5%);
* 4. Have measurable disease by International Myeloma Working Group (IMWG) criteria based on one or more of the following findings:

  * Serum M-protein≥ 1 g/dL（≥10 g/L）
  * Urine M-protein ≥ 200 mg/24 hour
  * Involved serum free light chain (FLCs) level≥10 mg/dL with FLCs abnormal ratio (<0.26或>1.65)
* 5. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1;
* 6. Diagnosis of MM with relapsed or refractory disease and have had at least 1 prior lines of therapy.

Exclusion Criteria:

* 1. Patients with plasmacytic leukemia or Waldenstrom's macroglobulinemia or POEMS syndrome (polyneuropathy, organ enlargement, endocrinopathy, monoclonal protein and skin lesions) or amyloidosis at screening;
* 2. Received any prior CAR-T therapy or BCMA targeted therapy;
* 3. Patients who have received autologous hematopoietic stem cell transplantation (ASCT) within 12 weeks prior to monocyte collection or history of allogeneic stem cell transplantation;
* 4. A history of immunodeficiency, including a positive HIV antibody test;
* 5. Hepatitis B surface antigen (HBsAg) positive and HBV-DNA above the lower limit of measurement or 1000 copies /mL (500 IU/mL), (whichever is lower), HCV antibody positive and HCV-RNA above the lower limit of measurement or 1000 copies /mL (whichever is lower);
* 6. Patients who, in the judgment of the investigator, need but are unable to receive prophylactic treatment for Pneumocystis, Herpes Simplex Virus (HSV), or Herpes Zoster (VZV) prior to initiation of treatment, or Syphilis confirmatory positive;
* 7. History of Bacillus Tuberculosis (TB) treatment within 2 years prior to first medication;
* 8. Patients with a history of interstitial lung disease and/or severe lung function impairment;
* 9. Have an active bacterial, fungal, or viral infection;
* 10.A history of severe cardiovascular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2032-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Up to approximately 6 months
  Incidence of adverse events (AEs)
Dose limiting toxicities (DLTs) | Up to 21 days
  Dose limiting toxicities (DLTs)

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to approximately 6 months
  Overall response rate (ORR)
Percentage of subjects who achieved complete response or strict complete response (CR/sCR) | Up to approximately 6 months
  Percentage of subjects who achieved complete response or strict complete response (CR/sCR)
Percentage of subjects who achieved very good partial response (VGPR) and higher response rate | Up to approximately 6 months
  Percentage of subjects who achieved very good partial response (VGPR) and higher response rate